CLINICAL TRIAL: NCT02407873
Title: Prognostic Impact of Frailty Assessed by Edmondon in Elderly Patient Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor of Anaesthesia and Intensive Care Medicine, University of Liege
Other Study IDs: 2013001
Record Dates: First submitted 2014-01-08; First posted 2015-04-03 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2015-10

CONDITIONS: Elective Cardiac Surgery
Keywords: aged of 75 years or more

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery
  Interventions: Other: Non

INTERVENTIONS:
Other: Non

SUMMARY:
The score on the Edmonton frail scale will be recorded in 250 consecutive patient aged of 75 years or more and undergoing elective cardiac surgery. In those patients the investigators will also record the ITU length of stay, the hospital length of stay, the incidence of complications, the ability to be discharged home and to live independently at postoperative day 30.

The ability of the Edmonton score to predict complication, prolonged hospital and ITU length of stay as well as loss of autonomy at discharge and day 30 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 75 yo and older
* Elective cardiac surgery

Exclusion Criteria:

* Refuse or inability to give consent
* Emergency surgery

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient aged 75 year and over undergoing elective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 Days

SECONDARY OUTCOMES:
Loss of autonomy at discharge (Edmonton score) | 30 Days
Loss of autonomy at day 30 (Edmonton score) | 30 days
Incidence of predefined complications | 30 Days
Length of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Liege, Liège, Belgium